CLINICAL TRIAL: NCT04376008
Title: Evaluation of Feasibility, Complications And Functional Results Of Free-Hand Transperineal Image Fusion Targeted Biopsies Under Local Anesthesia: A Prospective Study
Brief Title: A Prospective Study Of Free-Hand Transperineal Image Fusion Targeted Biopsies Under Local Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IUNU-PC-104
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PI-RADS 1-2 (Experimental): Standard prostate biopsy
  Interventions: Procedure: Standard prostate biopsy
- PI-RADS 3-5 (Experimental): Targeted and standard prostate biopsy
  Interventions: Procedure: Targeted and standard prostate biopsy

INTERVENTIONS:
Procedure: Standard prostate biopsy — Transperineal TRUS guided standard prostate biopsy (SB).
  Arms: PI-RADS 1-2
Procedure: Targeted and standard prostate biopsy — Transperineal Image fusion-guided targeted and standard prostate biopsy (TB+SB).
  Arms: PI-RADS 3-5

SUMMARY:
This trial aims to prospectively assess the feasibility, complications and functional results of free-hand transperineal image fusion targeted biopsies under local anesthesia in a large group of patients.

DETAILED DESCRIPTION:
12-core transrectal ultrasound (TRUS) biopsy is one of the most performed urological procedures and remains the standard method for prostate cancer (PCa) histological diagnosis according to the most recent Guidelines. During the last decade, the transperineal prostate biopsy has attracted renewed interest. However, only a few studies and no large prospective studies investigated complications of the transperineal approaches.

Image fusion of Multi-parameter MRI (mpMRI) and TRUS guided prostate targeted biopsy had equivalent results with standard 12-core biopsy. Combination of targeted and standard biopsy was recommended in recent Guidelines. Image fusion targeted biopsy needs satisfactory anesthetic effect, and no prospective studies investigated feasibility in this approach under local anesthesia.

The scientific urological community is focusing on detection rate and concordance with final pathology of the radical prostatectomy specimen, which remain the cornerstones to assess the accuracy of a prostate biopsy technique. In this study, the investigators will additionally assess the functional results of erectile function and urinary function.

Together, the investigators will perform free-hand image fusion targeted biopsies plus standard biopsies under local anesthesia in patients recruited in this study. Then, Feasibility, such as peri-procedural pain, changes in patients quality of life; complications, such as infection rate and bleeding rate; functional results, such as erectile function and urinary function; and concordance with final pathology will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men more than 18 years old with clinical suspicion of prostate cancer;
* Serum PSA ≤ 20 ng/ml within the previous 3 months;
* Suspected stage ≤ T2 on rectal examination (organ-confined prostate cancer) within the previous 3 months;
* No evidence of PSA increase by noncancerous factors, such as catheterization, bladder stones, or urinary tract infection including bacterial prostatitis;
* Able to provide written informed consent.

Exclusion Criteria:

* Prior prostate biopsy or prostate surgery;
* Prior treatment for prostate cancer;
* Contraindication to MRI (e.g. claustrophobia, pacemaker, estimated glomerular filtration rate ≤ 50mls/min);
* Contraindication to prostate biopsy.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Biopsy unfinished rates | 1 days
  The proportion of patients who failed to complete the biopsy due to various reasons during the biopsy
Pain score | 3 days peri-biopsy
  Numerical pain scale score during biopsy, the minimum to maximum value is 0 to 10, and higher scores mean a worse outcome
Hospitalization rate due to biopsy | 7 days post biopsy
  The proportion of subjects requiring hospitalization for various reasons within 7 days after puncture

SECONDARY OUTCOMES:
Detection rates of clinically significant PCa | 30 days post biopsy
  Clinically significant prostate cancer is considered as: biopsy Gleason score ≥3+4 or maximum cancer core length ≥5 mm.
Detection rates of PCa | 30 days post biopsy
  Prostate cancer is considered as: biopsy Gleason score ≥3+3
Biopsy-related complication rates | 30 days post biopsy
Biopsy time | 1 days
  How much time is used during biopsy
Consistency rate with final pathology | 30 days post biopsy
  Concordance rate between biopsy and final pathology
international index of erectile function-5 (IIEF-5) score | 30 days post biopsy
  pre- and post-procedural erectile function score, the minimum to maximum value is 0 to 25, and higher scores mean a better outcome
International prostate symptom score (IPSS) | 30 days post biopsy
  pre- and post-procedural urinary function score, the minimum to maximum value is 0 to 35, and higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China